CLINICAL TRIAL: NCT04616703
Title: Natural History of Benign Nonfunctioning Adrenal Tumors: 10 Year Follow-up Results
Brief Title: Natural History of NFAI: 10 Year Follow-up Results
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other); University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Principal Investigator, Mojca Jensterle, Clinical Professor, University Medical Centre Ljubljana
Other Study IDs: 00000
Record Dates: First submitted 2020-10-22; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Adrenal Incidentaloma
Keywords: adrenal incidentaloma; BMI; NFAI; MACE; long term follow up; natural history
MeSH Terms: conditions — Adrenal incidentaloma | interventions — Postmortem Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — venous blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BMI < 25 kg/m2: Those with NFAT and BMI < 25 kg/m2.
  Interventions: Radiation: CT imaging
- BMI 25-30 kg/m2: Those with NFAT and BMI 25-30 kg/m2.
  Interventions: Radiation: CT imaging
- BMI > 30 kg/m2: Those with NFAT and BMI > 30 kg/m2.
  Interventions: Radiation: CT imaging

INTERVENTIONS:
Radiation: CT imaging — CT of abdomen

SUMMARY:
The data on long term natural history of benign nonfunctioning adrenal tumors (NFATs) are lacking. The aim is to identify clinical characteristics associated with tumor growth and progression to mild autonomous cortisol excess over time.

DETAILED DESCRIPTION:
After being informed about the study, all patients with NFAT given written informed consent will underwent a control visit approximatly 10 years after initial visit at the outpateint clinic at the Department of Endocrinology, Diabetes and Metabolic Disease, University Medical Center Ljubljana, Ljubljana, Slovenia. The included patients will be divided in three groups regarding the BMI as follows: BMI < 25 kg/m2, 25-30 kg/m2 and > 30 kg/m2. The investigators will assess clinical, and laboratory parameters and CT findings at the follow up visit and compere them to baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

- Patients hospitalized because of NFAI between 2005-2012 at the Department of Endocrinology, Diabetes and Metabolic Disease, University Medical Center Ljubljana, Ljubljana, Slovenia.

Exclusion Criteria:

* age below 18 years
* relatives reported that patient died in the time since hospitalization
* patient did not want a follow up
* patient did not attend follow up appointment
* patient underwent adrenalectomy
* misdiagnosis / missing main information in hospitalization record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with diagnosisi of NFAI, hospitalized between 2005-2012 at the Department of Endocrinology, Diabetes and Metabolic Disease, University Medical Center Ljubljana, Ljubljana, Slovenia.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Natural History of NFAT - horomnal activity | 10 years
  To determine if and in how many pateints NFAI progressed to MACE.
  NFAI: when cortisol after 1 mg overnight dexamethasone (ODST) suppression test is < 50 nmol/l and no typical clinical signs of Cushing's syndrome are present. Pheochromocytoma and primary aldosteronism will be excluded.
  MACE: when cortisol after 1 mg overnight dexamethasone (ODST) suppression test is > 50 nmol/l.
Natural History of NFAT - growth | 10 years
  To determine the change in size of NFAI on the CT scan (mm).
Natural History of NFAT - BMI | 10 years
  To determine the change in BMI and its correlation with outcome 1 and 2.
  Weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Mojca Jensterle, MD, PhD, Study Director — University Medical Center Ljubljana, Slovenia
Locations (1):
- Department of Internal Medicine, Faculty of Medicine, University of Ljubljana, Ljubljana, Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No